CLINICAL TRIAL: NCT06377397
Title: Selective Antibiotics When Symptoms Develop Versus Universal Antibiotics for Preterm Neonates At-risk of Early-onset Bacterial Sepsis: a Multicentric, Randomized, Controlled, Non-inferiority Trial (the SAUNA Trial)
Brief Title: Selective Antibiotics When Symptoms Develop Versus Universal Antibiotics for Preterm Neonates
Acronym: SAUNA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Indian Council of Medical Research (Other Government)
Collaborators: Lady Hardinge Medical College (Other Government); King George's Medical University (Other); Indira Gandhi Institute of Child Health (Unknown); Institute of Obstetrics and Gynecology (Unknown); Government Medical College, Chandigarh (Other); Pandit Bhagwat Dayal Sharma, PGIMS, Rohtak (Other); Government Medical College, Aurangabad (Other Government); King Edward Memorial Hospital, Mumbai (Other Government)
Responsible Party: Principal Investigator, Sourabh Dutta, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIRPIG-2023-0000070
Record Dates: First submitted 2024-03-26; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Sepsis; PROM, Preterm (Pregnancy); Early-Onset Neonatal Sepsis; Preterm Premature Rupture of Membrane; Preterm Birth
Keywords: Prolonged rupture of membranes; Preterm premature rupture of membranes; Early-onset neonatal sepsis; Selective antibiotics; Non-inferiority trial
MeSH Terms: conditions — Sepsis; Fetal Membranes, Premature Rupture; Neonatal Sepsis; Preterm Premature Rupture of the Membranes; Premature Birth | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Neonates will be randomized to 1 of the following groups:
  1. Group 1: Intervention group (Selective antibiotic group)
  2. Group 2: Comparison group (Universal antibiotic group)
Who Masked: Outcomes Assessor
Masking Description: Project staff, nurses and resident doctors looking after the neonate will not be blinded. The assessment of the primary outcome will be performed by a blinded adjudicator, who is not involved in the recruitment and monitoring of subjects. A part of the case report form (CRF) containing relevant details of all episodes of sickness in the 1st week of life will be detached from the main form and will be sent to the blinded adjudicator. This part will be linked to the main form only by a unique identification number. No patient identifiers or allocation group will be mentioned on the part sent to the blinded adjudicator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective antibiotic group (Experimental): Antibiotics will be administered selectively to a subset of at-risk neonates who develop clinical signs of sepsis.
  Interventions: Drug: Antibiotics
- Comparison group (Active Comparator): Antibiotics will be pre-emptively administered to all neonates at risk of sepsis.
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Antibiotics — In experimental arm, intravenous antibiotics as per the written down empirical antibody policy of the unit will be administered selectively to those newborn infants who later develop clinical signs of sepsis according to a predefined repertory of clinical signs.
  In active comparator arm, intravenous antibiotics as per the written down empirical antibody policy of the unit will be administered pre-emptively to all newborn infants from enrollment even if they do not have any clinical signs of sepsis at enrollment
  Other Names: Intravenous antibiotics as per written down empirical antibiotic policy of the unit

SUMMARY:
Preterm infants are born at less than 37 weeks of pregnancy. Sometimes a break or tear in the fluid filled bag that surrounds and protects the infant during pregnancy leads to an untimely birth. This state puts the infant at risk of serious condition called sepsis. Sepsis is a condition in which body responds inappropriately to an infection. Sepsis may progress to septic shock which can result in the loss of life. Doctors give antibiotics to treat sepsis.

The goal of this research study is to find out:

1. Among neonates at risk of early-onset neonatal sepsis, whether a policy of administering antibiotics selectively to a subset of at-risk infants who later develop signs of sepsis is not inferior to administering antibiotics to all at-risk infants in the 1st week of life.
2. To find out if infants receiving selective antibiotics (as above) compared to those receiving antibiotics from birth (as above) require fewer antibiotic courses of 48 hours duration or more in the 1st week of life.
3. To find out whether infants receiving selective antibiotics (as above) compared to those receiving antibiotics from birth (as above) are significantly different with respect to a wide range of secondary outcomes (listed under "Outcomes").

DETAILED DESCRIPTION:
Sepsis is the major cause of neonatal mortality and early-onset neonatal sepsis (EONS) accounts for more than two-thirds of all cases of neonatal sepsis. Prolonged rupture of membranes (PROM) and preterm premature rupture of membranes (pPROM) are important risk factors of EONS. There is equipoise in the published literature whether antibiotics must be immediately initiated among all preterm neonates (<35 weeks gestation) delivered following PROM or pPROM who are asymptomatic at birth or whether antibiotics can be selectively administered if and when the at-risk neonates become symptomatic.

Among neonates <35 weeks gestation born with PROM >18 hours or pPROM and who are either asymptomatic or have no symptoms of sepsis at 4 hrs postnatally (P), is selectively administering antibiotics to neonates who later develop clinical sepsis [I] compared to administering antibiotics pre-emptively to all at-risk neonates [C] non-inferior with respect to the composite outcome of "mortality and/or culture-positive sepsis and/or severe sepsis" [O] within 7 days after enrolment [T] by an absolute margin of 7% [E] in a randomized controlled trial (S)? The trial will also have a superiority outcome: "need for antibiotic treatment lasting greater than 48 hours within 7 days after enrolment". The absolute superiority margin will be 50%.

The main objectives are as follows:

1. To determine whether antibiotics administered selectively to at-risk preterm neonates [<35 weeks gestation with prolonged rupture of membranes (PROM) or preterm premature rupture of membranes (pPROM)] when they develop signs of sepsis compared to administering antibiotics from birth to all at-risk neonates is non-inferior with respect to the primary outcome of "mortality or any episode of culture-positive sepsis or severe sepsis" in the 1st week of life
2. To determine whether neonates receiving selective antibiotics (as above) compared to those receiving antibiotics from birth (as above) are superior with respect to the co-primary outcome of fewer antibiotic courses of 48 hours duration or more in the 1st week of life
3. To determine whether neonates receiving selective antibiotics (as above) compared to those receiving antibiotics from birth (as above) are significantly different with respect to a wide range of secondary outcomes (listed under "Outcomes")

ELIGIBILITY:
Inclusion criteria:

* Gestational age of 26 to 34 weeks
* Chronological age 4 hours
* Have any one or both of the following risk factors of EONS:

  * Prolonged rupture of membranes >18 hours
  * Pre-labour rupture of membranes [as all subjects will be preterm, this is effectively pPROM]
* Are either asymptomatic or have no signs attributable to sepsis at 4 hours. This will be defined as absence of the following clinical signs or need for interventions mentioned below:

  1. Apnea (Standard definition) requiring intervention at any time until enrolment.
  2. Need for a fluid bolus or inotropic support at any time until enrolment.
  3. Seizures or seizure-like activity at any time until enrolment.
  4. Upper GI bleed in the absence of a history of ante-partum hemorrhage at any time until enrolment.
  5. Pus from any site at any time until enrolment.
  6. Need for CPAP >6 cms of water with FiO2 >35% at 6-8 hours OR need for CPAP £6 cms and FiO2 £35% but with increasing requirement of support**
  7. Chest Xray (if performed) with radiological features of pneumonia.
  8. Need for intubation and mechanical ventilation.
  9. Temperature >37.5°C or <36°C, unexplained by environmental causes
  10. Feed intolerance [bilious or bloodstained vomiting (or gastric residuals) or visibly distended abdomen or >50% of the previous feed volume as gastric residuals]
  11. Lethargy or unarousability
  12. Sclerema

      Exclusion Criteria:

      Subjects will be excluded if they have any 1 of the following:

  <!-- -->

  1. Life-threatening congenital malformation
  2. Severe perinatal asphyxia (Apgar score <5 at 10 minutes or cord pH <7.0)
  3. Clinical chorioamnionitis# [see definition below]
  4. Foul-smelling liquor
  5. Multiple gestation
  6. Received a dose of antibiotics
  7. Positive amniotic fluid culture (if performed and available prior to randomization)
  8. Treating neonatologist unwilling to enroll the patient in the trial on the grounds that the patient needs antibiotics.

     -

Ages: 0 Hours to 4 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2028-04-14 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality and/or any episode of culture-positive sepsis and/or severe sepsis* within the 1st 7 days after randomization | Within 1st 7 days after randomization
  Either mortality due to any cause and/or an episode of culture-positive sepsis and/or severe sepsis. These outcomes will be measured within the "1st 7 days after randomization", which for all practical purposes, is equivalent to the "1st 7 days of life" since participants will be randomized at about 4 hours of life. Hence, the duration expressed after randomization and of life will be used interchangeably for this outcome and other outcomes.
Need for intravenous antibiotics for ≥ 48 hours within the 1st 7 days after randomization | Within 1st 7 days after randomization
  Requirement for intravenous antibiotic courses whose duration is ≥ 48 hours with the onset of the course within the first 7 days after randomization. For all practical purposes, this would be equivalent to the 1st 7 days of life since participants will be randomized at about 4 hours of life.

SECONDARY OUTCOMES:
All-cause Mortality within 1st 7 days after randomization | During 1st 7 days after randomization
  Mortality due to any cause
Blood culture-positive sepsis of any severity within 1st 7 days after randomization | Within 1st 7 days after randomization
  Blood culture proven septicemia
Episode of severe sepsis within 1st 7 days after randomization | Within 1st 7 days after randomization
  Any episode of severe sepsis during 1st 7 days after randomization. Severe sepsis be defined as clinical signs of sepsis AND either a positive blood culture or laboratory evidence of sepsis (either CRP OR Procalcitonin above the age-appropriate cut-off value OR any two of the CBC parameters outside the age-appropriate ranges OR chest x-ray suggestive of pneumonia) AND one or more of the following indices of severity [Need for intubation and mechanical ventilation, Need for inotropes >10 mic/kg/min dopamine or >10 mic/kg/min dobutamine or adrenaline > 0.05 mic/kg/min, Need for exchange transfusion, Need for platelet concentrates or FFP, Meningitis (defined as either CSF culture positive or Gram stain positive or Cell count >25/microlitre or glucose <25 mg/dl or protein >180 mg/dl)]
Composite of mortality/blood culture positive sepsis/severe sepsis within 1st 72 hours after randomization | Within first 72 hour after randomization
  Either mortality and/or blood culture-positive sepsis and/or severe sepsis
Individual components of composite outcome within 1st 72 hours after randomization | Within 1st 72 hours after randomization
  Separately mortality, blood culture-positive sepsis or severe sepsis
Composite of mortality/blood culture positive sepsis/severe sepsis during hospital stay | During hospital stay upto 100 days after randomization
  Either mortality due to any cause and/or blood culture-positive sepsis and/or severe sepsis during hospital stay, with maximum duration of observation during hospital stay being capped at 100 days
Individual components of composite outcome during hospital stay | During hospital stay upto 100 days after randomization
  Separately mortality, blood culture-positive sepsis or severe sepsis during hospital stay, with maximum duration of observation during hospital stay being capped at 100 days
Necrotizing enterocolitis, stage II-III by modified Bell's staging criteria during hospital stay | During hospital stay upto 100 days after randomization
  Necrotizing enterocolitis stage II-III by modified Bell's staging criteria during hospital stay, with maximum duration of observation during hospital stay being capped at 100 days after randomization
Composite of mortality/blood culture positive sepsis/severe sepsis during 1st 30 days after randomization | During 1st 30 days after randomization
  Either all-cause mortality and/or blood culture-positive sepsis and/or severe sepsis during the 1st 30 days after randomization
Individual components of composite outcome during 1st 30 days | During 1st 30 days after randomization
  Separately, all-cause mortality, blood culture-positive sepsis or severe sepsis during the 1st 30 days after randomization
Necrotizing enterocolitis, stage II-III by modified Bell's staging criteria | During 1st 30 days after randomization
  Necrotizing enterocolitis, stage II-III by modified Bell's staging criteria during the 1st 30 days after randomization
Sepsis-related mortality within 1st 72 hours after randomization | Within 1st 72 hours after randomization
  Mortality due to sepsis within 1st 72 hours. The decision of the treating team will be recorded for attributing mortality to sepsis.
Sepsis-related mortality within 7 day after randomization | Within 7 days after randomization
  Mortality due to sepsis within 7 days after randomization. The decision of the treating team will be recorded for attributing mortality to sepsis.
Sepsis-related mortality during hospital stay after randomization | During hospital stay upto 100 days after randomization
  Mortality due to sepsis during hospital stay. The decision of the treating team will be recorded for attributing mortality to sepsis.
Sepsis-related mortality during 1st 30 days after randomization | During 1st 30 days after randomization
  Mortality due to sepsis during 1st 30 days after randomization
Clinical sepsis within 1st 72 hours after randomization | Within 1st 72 hours after randomization
  Episodes of clinical EONS (as per definition from a repertoire of clinical signs with normal lab parameters) within 1st 72 hours
Clinical sepsis within 7 days after randomization | Within 7 days after randomization
  Episodes of clinical EONS (as per definition from a repertoire of clinical signs with normal lab parameters) within 7 days
Clinical sepsis during hospital stay | During hospital stay upto 100 days
  Episodes of clinical EONS (as per definition from a repertoire of clinical signs with normal lab parameters) during hospital stay, with maximum duration of observation during hospital stay being capped at 100 days after randomization
Clinical sepsis within 1st 30 days after randomization | During 1st 30 days after randomization
  Episodes of clinical EONS (as per definition from a repertoire of clinical signs with normal lab parameters) within 1st 30 days of life
Episode of Probable EONS within 72 hours after randomization | Within 72 hours after randomization
  Episode of Probable EONS [as per definition from a repertoire of clinical signs, AND with abnormal age-appropriate values of one or more of TLC, ANC, CRP, PCT, chest x-ray suggestive of pneumonia AND with sterile blood culture]
Episode of Probable EONS within 7 days after randomization | Within 7 days after randomization
  Episode of Probable EONS [as per definition from a repertoire of clinical signs, AND with abnormal age-appropriate values of one or more of TLC, ANC, CRP, PCT, chest x-ray suggestive of pneumonia AND with sterile blood culture]
Episode of asymptomatic proven EONS within 72 hours after randomization | Within 72 hours after randomization
  Episode of asymptomatic proven EONS [asymptomatic but baseline blood culture positive with non-contaminant organism]
Need for sepsis workup during 1st 72 hours after randomization | During 1st 72 hours after randomization
  ["Sepsis workup" defined as one or more of CBC, CRP, Procalcitonin, blood culture] during 1st 72 hours of life
Need for sepsis workup during 1st 7 days after randomization | During 1st 7 days after randomization
  "Sepsis workup" defined as one or more of CBC, CRP, Procalcitonin, blood culture during 1st 7 days of life
Need for sepsis workup during 1st 30 days after randomization | During 1st 30 days after randomization
  "Sepsis workup" defined as one or more of CBC, CRP, Procalcitonin, blood culture during 1st 30 days of life
Need for sepsis workup during hospital stay | During hospital stay upto 100 days
  "Sepsis workup" defined as one or more of CBC, CRP, Procalcitonin, blood culture during hospital stay, with the period of observation during hospital stay being capped at 100 days
Cumulative duration of antibiotic therapy during 1st 7 days after randomization | During 1st 7 days after randomization
  Cumulative duration of antibiotic therapy during the 1st 7 days, which may include the sum of the durations of multiple courses of antibiotics, either in continuation or discontinuous. If any course of antibiotics continues beyond the 1st 7 days after randomization, only that portion of the antibiotic course would be included until the 1st 7 days after randomization.
Cumulative duration of antibiotic therapy during 1st 72 hrs after randomization | During 1st 72 hours after randomization
  Cumulative measure of antibiotics therapy during the 1st 72 hours
Cumulative duration of antibiotic therapy during hospital stay | During hospital stay upto 100 days after randomization
  Cumulative measure of antibiotics therapy during hospital stay, with the period of observation during hospital stay capped at 100 days
Duration of hospitalization | Upto 100 days
  Full length of hospital stay, with the period capped at 100 days
Episodes of healthcare associated infection during hospital stay. | From after 72 hours until 100 days during hospital stay
  Defined as any episode of culture positive sepsis with onset after 72 hours of life or any episode of culture-positive sepsis if baseline blood culture was sterile, with the period of observation during hospital stay capped at 100 days
Adverse effects until day 30 after randomization | During 30 days after randomization
  Adverse effects will be recorded as per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Serious adverse effects until day 30 after randomization | During 30 days after randomization
  Serious adverse effects will be recorded as per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Sourabh Dutta, MD, Ph.D, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
Anonymized, individual patient data pertaining to publications from the study which are in the public domain will be shared with other researchers planning to conduct a study, upon reasonable written request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available one year after the publication from the study for a period of 3 years
Access Criteria: To be decided

REFERENCES:
- [Result] Sankar MJ, Neogi SB, Sharma J, Chauhan M, Srivastava R, Prabhakar PK, Khera A, Kumar R, Zodpey S, Paul VK. State of newborn health in India. J Perinatol. 2016 Dec;36(s3):S3-S8. doi: 10.1038/jp.2016.183. PMID 27924104
- [Result] Lawn JE, Blencowe H, Oza S, You D, Lee AC, Waiswa P, Lalli M, Bhutta Z, Barros AJ, Christian P, Mathers C, Cousens SN; Lancet Every Newborn Study Group. Every Newborn: progress, priorities, and potential beyond survival. Lancet. 2014 Jul 12;384(9938):189-205. doi: 10.1016/S0140-6736(14)60496-7. Epub 2014 May 19. PMID 24853593
- [Result] Chaurasia S, Sivanandan S, Agarwal R, Ellis S, Sharland M, Sankar MJ. Neonatal sepsis in South Asia: huge burden and spiralling antimicrobial resistance. BMJ. 2019 Jan 22;364:k5314. doi: 10.1136/bmj.k5314. PMID 30670451
- [Result] Chan GJ, Lee AC, Baqui AH, Tan J, Black RE. Risk of early-onset neonatal infection with maternal infection or colonization: a global systematic review and meta-analysis. PLoS Med. 2013 Aug;10(8):e1001502. doi: 10.1371/journal.pmed.1001502. Epub 2013 Aug 20. PMID 23976885
- [Result] Puopolo KM, Benitz WE, Zaoutis TE; COMMITTEE ON FETUS AND NEWBORN; COMMITTEE ON INFECTIOUS DISEASES. Management of Neonates Born at >/=35 0/7 Weeks' Gestation With Suspected or Proven Early-Onset Bacterial Sepsis. Pediatrics. 2018 Dec;142(6):e20182894. doi: 10.1542/peds.2018-2894. PMID 30455342
- [Result] Wolf RL, Olinsky A. Prolonged rupture of fetal membranes and neonatal infections. S Afr Med J. 1976 Apr 3;50(15):574-6. PMID 772827
- [Result] Berardi A, Fornaciari S, Rossi C, Patianna V, Bacchi Reggiani ML, Ferrari F, Neri I, Ferrari F. Safety of physical examination alone for managing well-appearing neonates >/= 35 weeks' gestation at risk for early-onset sepsis. J Matern Fetal Neonatal Med. 2015 Jul;28(10):1123-7. doi: 10.3109/14767058.2014.946499. Epub 2014 Sep 10. PMID 25034325
- [Result] Berardi A, Buffagni AM, Rossi C, Vaccina E, Cattelani C, Gambini L, Baccilieri F, Varioli F, Ferrari F. Serial physical examinations, a simple and reliable tool for managing neonates at risk for early-onset sepsis. World J Clin Pediatr. 2016 Nov 8;5(4):358-364. doi: 10.5409/wjcp.v5.i4.358. eCollection 2016 Nov 8. PMID 27872823
- [Result] Berardi A, Spada C, Reggiani MLB, Creti R, Baroni L, Capretti MG, Ciccia M, Fiorini V, Gambini L, Gargano G, Papa I, Piccinini G, Rizzo V, Sandri F, Lucaccioni L; GBS Prevention Working Group of Emilia-Romagna. Group B Streptococcus early-onset disease and observation of well-appearing newborns. PLoS One. 2019 Mar 20;14(3):e0212784. doi: 10.1371/journal.pone.0212784. eCollection 2019. PMID 30893310
- [Result] Cantoni L, Ronfani L, Da Riol R, Demarini S; Perinatal Study Group of the Region Friuli-Venezia Giulia. Physical examination instead of laboratory tests for most infants born to mothers colonized with group B Streptococcus: support for the Centers for Disease Control and Prevention's 2010 recommendations. J Pediatr. 2013 Aug;163(2):568-73. doi: 10.1016/j.jpeds.2013.01.034. Epub 2013 Mar 8. PMID 23477995
- [Result] Joshi NS, Gupta A, Allan JM, Cohen RS, Aby JL, Weldon B, Kim JL, Benitz WE, Frymoyer A. Clinical Monitoring of Well-Appearing Infants Born to Mothers With Chorioamnionitis. Pediatrics. 2018 Apr;141(4):e20172056. doi: 10.1542/peds.2017-2056. PMID 29599112
- [Result] Chiruvolu A, Petrey B, Stanzo KC, Daoud Y. An Institutional Approach to the Management of Asymptomatic Chorioamnionitis-Exposed Infants Born >/=35 Weeks Gestation. Pediatr Qual Saf. 2019 Dec 5;4(6):e238. doi: 10.1097/pq9.0000000000000238. eCollection 2019 Nov-Dec. PMID 32010864
- [Result] Investigators of the Delhi Neonatal Infection Study (DeNIS) collaboration. Characterisation and antimicrobial resistance of sepsis pathogens in neonates born in tertiary care centres in Delhi, India: a cohort study. Lancet Glob Health. 2016 Oct;4(10):e752-60. doi: 10.1016/S2214-109X(16)30148-6. PMID 27633433

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT06377397/Prot_SAP_000.pdf